CLINICAL TRIAL: NCT00550706
Title: Drug Utilization Prevalence in a Pediatric Care Medical Center
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: PDU2724_CTIL
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Infectious Diseases; Metabolic Diseases; Cancer
Keywords: Prescription point prevalence; Drug utilization; Define Daily Dose
MeSH Terms: conditions — Communicable Diseases; Metabolic Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1Pediatric Dept A: Children's files from this department will be analysed once weekly and medication prescription data will be registered
- 2 Pediatric Dept B: Children's files from this department will be analysed once weekly and medication prescription data will be registered

SUMMARY:
One year prospective analysis of drug utilization and prescription point prevalence of medications in a pediatric tertiary care university medical center. Off-label use of medications in the study population will be also registered.

ELIGIBILITY:
Inclusion Criteria:

* All admitted children receiving at least one prescribed or OTC medication.

Exclusion Criteria:

* All admitted children who do not get a prescribed or OTC medication.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Admitted children for medical treatment in two different pediatric departments
Sampling Method: Non-Probability Sample
Enrollment: 567 (Actual)
Dates: Start 2007-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Descriptive use of medications | One year

CONTACTS AND LOCATIONS:
Overall Officials: Norberto Krivoy, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel